CLINICAL TRIAL: NCT03339544
Title: Effect of Celebrex Pre-medication on the Intra and Post-treatment Endodontic Pain in Teeth With Symptomatic Irreversible Pulpitis: Double Blind Randomized Clinical Trial
Brief Title: Celebrex Premedication in Teeth With Symptomatic Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yousra Khaled Mohamed Ezzat, Resident at Endodontic department. Faculty of Oral and Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: celebrex premedication
Record Dates: First submitted 2017-11-01; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celebrex premedication (Experimental): Celebrex is a NSAID with selective COX-2 inhibition properties, is given as an intervention to assess the pain
  Interventions: Drug: Celebrex premedication
- Placebo tablets (Placebo Comparator): placebo tablets to compare the efficacy of Celebrex on the intra-operative and post-operative pain accompanying endodontic treatment of teeth with irreversible pulpits
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celebrex premedication — celebrex (celecoxib) 200mg is a non-steroidal anti-infalmmatory drug with selective COX-2 inhibition.
  Other Names: Celecoxib
  Arms: Celebrex premedication
Drug: Placebo — placebo is given as a tablet before initiation of endodontic treatment
  Arms: Placebo tablets

SUMMARY:
Assessing the efficacy of Celebrex premedication on pain during and after endodontic treatment in teeth with symptomatic irreversible pulpits

DETAILED DESCRIPTION:
Owing to the painful nature of endodotnic treatment in teeth with irreversible pulpits, administration of an analgesic and anti-inflammatory could help to lessen the perception of pain, hence decreasing the patient apprehension.

Previous clinical trials have shown that the use of NSAIDS as a premedication prior to endodontic treatment was effective in reducing the pain and increasing the anesthetic success, since as high as 80% of the patients with pre-operative pain experience pain after endodontic treatment.

In this study, Celebrex (Celecoxib) 200mg will be given to the patients 1 hour before initiation of the treatment, and its effect on reducing the pain will be compared with a placebo.

Celebrex being a selective COX-2 inhibitor, it will spare the physiological tissue prostaglandin production while inhibiting the inflammatory prostaglandin production thus allow for effective analgesia with fewer side effects than Non-Selective NSAIDS (nsNSAIDS).

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients
* Patients able to understand Visual Analogue Scale and sign the informed conset

Mandibular molar teeth with:

* Preoperative sharp pain
* Vital pulp tissue
* Normal peripaical radiographic appearance or slight widening of the lamina dura

Exclusion Criteria:

* Patients allergic to NSAIDS
* Pregnant females
* Patients having significant systemic disorder
* Patients with psychological disturbances
* Patients with bruxism or clenching

Teeth that have:

* Associated with swelling or fistulous tract
* Acute or chronic periapical abscess
* Greater than grade I mobility
* Periodontitis
* No possible restorability
* previous endodontic treatment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
pain intensity (intra-operative pain) | 1 hour after administration of the drug up to 2 hours till the end of endodontic treatment
  pain intensity during endodontic treatment, measured by Visual Analogue Scale (pain scale)

SECONDARY OUTCOMES:
alleviation of pain severity | 24 hours
  severity of pain is measured by Visual Analogue Scale
number of analgesic tablets taken by the patient after endodontic treatment | 24 hours
  counting the number of analgesic tablets taken by the patient after the treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee Y, Rodriguez C, Dionne RA. The role of COX-2 in acute pain and the use of selective COX-2 inhibitors for acute pain relief. Curr Pharm Des. 2005;11(14):1737-55. doi: 10.2174/1381612053764896. PMID 15892672
- [Result] Lapidus D, Goldberg J, Hobbs EH, Ram S, Clark GT, Enciso R. Effect of premedication to provide analgesia as a supplement to inferior alveolar nerve block in patients with irreversible pulpitis. J Am Dent Assoc. 2016 Jun;147(6):427-37. doi: 10.1016/j.adaj.2016.01.006. Epub 2016 Mar 4. PMID 26952243